CLINICAL TRIAL: NCT03172221
Title: Clinical Performance of the Histidine Rich Protein 2 (HRP2) Highly Sensitive Rapid Diagnostic Test (HS-RDT) for Malaria Diagnosis in Pregnant Women
Brief Title: Clinical Performance of the HRP2 HS-RDT for Malaria Diagnosis in Pregnant Women
Acronym: HSRDT MiP
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Other Study IDs: 7815-2/1
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Plasmodium Falciparum; Pregnancy Malaria; Diagnoses Disease
Keywords: malaria; pregnancy; diagnosis; low-transmission; Plasmodium falciparum; rapid diagnostic test
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HS-RDT — A single finger-prick blood sample will be collected and used to test participants with the HS-RDT. The results of the results of the test will not be used for treatment purposes nor used to inform patient care.
  Other Names: ultrasensitive RDT

SUMMARY:
This is a cross-sectional and multicentre clinical trial to study the performance of the Histidine Rich Protein 2 (HRP2) highly sensitive rapid diagnostic test (HS-RDT) for the detection of malaria during pregnancy in low transmission settings from Colombia and Indonesia. The new HS-RDT will be compared with conventional good quality RDTs, microscopy, and NAATs [loop-mediated isothermal amplification (LAMP), nested PCR (nPCR)], in peripheral blood samples with quantitative reverse transcription PCR (qRT-PCR) as reference standard.

DETAILED DESCRIPTION:
The activities proposed will be performed in the context of health centres receiving pregnant women for antenatal care visit. Finger-prick blood (300 µL) will be collected and used to test for malaria with the HS-RDT, as well as with conventional good quality RDTs, microscopy and local NAATs (LAMP and nPCR). Dried blood spots will also be collected for qRT-PCR testing. Patient information (demographics, obstetric history, malaria prevention measures, etc.) as well as laboratory results will be recorded and entered into a dedicated database.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed pregnancy and registered to the antenatal care programme in the local health centre
* Resident for at least 1 year in the study site
* Age ≥ 15
* Accepting to participate with willingness to give informed consent (pregnant adolescents younger than 18 y/o (age < 18) will be considered only if they are accompanied by parent or carer if it is requested by local Institutional Review Boards)
* Willingness to provide finger-prick blood sample at enrolment

Exclusion Criteria:

* Past history of malaria and/or antimalarial drugs in the last three months
* Positive for malaria by microscopy and conventional RDT testing in any previous study screening visit
* Presence of severe malaria as defined by WHO guidelines at the moment of recruitment
* Presence of symptoms and signs of other severe disease and central nervous system infections, as defined by WHO guidelines.

Min Age: 15 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study will include pregnant women
Study Population: Consecutive pregnant women self-presenting at the selected health care facilities and meeting the eligibility criteria will be invited to participate in the study. After study staff provides full information about the study, pregnant women willing to participate will be asked to sign the informed consent form. They will consent to be interviewed and to provide finger-prick blood. For women younger than 18 years old, additional approval from the parent or legal guardian will be needed if required by local Institutional Review Board (IRB). Participants will be invited to participate at any visit at any trimester.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  Sensitivity, specificity, negative predictive value, positive predictive value, diagnostic odds ratio (DOR) and the area under the receiver operating characteristic curve (AUROC) of HRP2 HS-RDT for the detection of P. falciparum during pregnancy, compared with conventional good quality RDTs, microscopy and NAATs (LAMP, nPCR,), in peripheral blood with qRT-PCR as reference standard.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Centro de Salud el Reposo, Quibdó
  - Hospital Divino Nino, Tumaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasquez AM, Velez G, Medina A, Serra-Casas E, Campillo A, Gonzalez IJ, Murphy SC, Seilie AM, Ding XC, Tobon Castano A. Evaluation of highly sensitive diagnostic tools for the detection of P. falciparum in pregnant women attending antenatal care visits in Colombia. BMC Pregnancy Childbirth. 2020 Jul 31;20(1):440. doi: 10.1186/s12884-020-03114-4. PMID 32736543